CLINICAL TRIAL: NCT02712008
Title: A Randomized, Double-Masked, Active-Controlled, Phase 2 Study of the Efficacy, Safety, and Tolerability of Repeated Doses of Intravitreal REGN910-3 in Patients With Diabetic Macular Edema
Brief Title: Anti-vasculaR Endothelial Growth Factor plUs Anti-angiopoietin 2 in Fixed comBination therapY: Evaluation for the Treatment of Diabetic Macular Edema
Acronym: RUBY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R910-3-DME-1518
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- REGN910-3 (3 mg: 2 mg) (Experimental): Participants were administered intravitreal injection of REGN910-3 (3 milligram (mg):2 mg) every 4 weeks (Q4) on Day 1, Week 4, and Week 8 for 3 initial doses followed by every Week 8 (Q8) dosing beginning at Week 16 up to Week 32.
  Interventions: Drug: REGN910-3
- REGN910-3 (6 mg:2 mg) (Experimental): Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to week 12.
  Interventions: Drug: REGN910-3
- Aflibercept 2 mg (Active Comparator): Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)
- REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 (Experimental): Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) at Week 16 and Q8 through Week 32.
  Interventions: Drug: REGN910-3
- REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 (Experimental): Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) at Week 20 and Q12 through Week 32.
  Interventions: Drug: REGN910-3
- Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 (Experimental): Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI at Week16 and Q8 through Week 32.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)
- Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 (Experimental): Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI at Week 20 and Q12 through Week 32.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI)
- Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8 (Experimental): Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) at week 16 and Q8 through week 32.
  Interventions: Drug: REGN910-3; Drug: Intravitreal Aflibercept Injection (IAI)

INTERVENTIONS:
Drug: REGN910-3 — Co-formulation for intravitreal (IVT) injection consisting of REGN910 (nesvacumab) and REGN3 (aflibercept)
  Arms: Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; REGN910-3 (3 mg: 2 mg); REGN910-3 (6 mg:2 mg); REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8
Drug: Intravitreal Aflibercept Injection (IAI)
  Other Names: EYLEA® (aflibercept) Injection; BAY86-5321
  Arms: Aflibercept 2 mg; Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8

SUMMARY:
The primary objective of the study was to compare the efficacy of intravitreal (IVT)-administered REGN910-3 compared to intravitreal aflibercept injection (IAI) in improving best corrected visual acuity (BCVA) in participants with diabetic macular edema (DME).

ELIGIBILITY:
Key Inclusion Criteria:

1. Men or women ≥18 years of age with type 1 or type 2 diabetes mellitus who have clinically significant DME with central involvement in the study eye
2. BCVA ETDRS letter score of 73 to 24 (Snellen equivalent of 20/40 to 20/320) in the study eye
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Key Exclusion Criteria:

1. Evidence of macular edema due to any cause other than diabetes mellitus in either eye
2. IVT anti-VEGF in the study eye within 12 weeks of the screening visit
3. Panretinal laser photocoagulation or macular laser photocoagulation in the study eye within 3 months of screening

Note: Other inclusion/ exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2016-03-02; Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (51):
- United States (51):
  - Mesa, Arizona
  - Tucson, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Mountain View, California
  - Oceanside, California
  - Palm Desert, California
  - Colorado Springs, Colorado
  - New London, Connecticut
  - Lakeland, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - ‘Aiea, Hawaii
  - Chicago, Illinois
  - New Albany, Indiana
  - Shawnee Mission, Kansas
  - Lexington, Kentucky
  - Portland, Maine
  - Baltimore, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Minneapolis, Minnesota
  - Florissant, Missouri
  - Las Vegas, Nevada
  - Bloomfield, New Jersey
  - Edison, New Jersey
  - Teaneck, New Jersey
  - Albany, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Kingston, Pennsylvania
  - Florence, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Harlingen, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Willow Park, Texas
  - Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 70 sites in US. A total of 438 participants were screened in the study.
Pre-assignment Details: Out of 438 participants, 302 were randomized & treated in study. Participants were randomized in 1:2:3 to receive REGN910-3 3:2mg, REGN910-3 6:2mg & 2mg intravitreal aflibercept injection followed by re-randomization at week 12 in REGN910-3 6:2mg & IAI 2mg arm. Not all participants who completed Week 12 were re-randomized & continued to Week 36.
Groups:
- REGN910-3 (3 mg: 2 mg): Participants were administered intravitreal injection of REGN910-3 (3 milligram [mg]:2 mg) every 4 weeks (Q4) on Day 1, Week 4, and Week 8 for 3 initial doses followed by every Week 8 (Q8) dosing beginning at Week 16 up to Week 32.
- Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At week 12, participants were re-randomized to receive IAI at week 16 and Q8 through week 32.
Period: Baseline (Day 1) up to Week 12
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Started | 50 | 100 | 152 | 0 | 0 | 0 | 0 | 0
Completed | 46 | 97 | 148 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other Unspecified | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: From Week 12 up to Week 36
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Started | 45 (Out of 46 participants that completed Week 12, 45 re-randomized for treatment from Week 12 to 36) | 0 (Out of 97 participants that completed Week 12, 96 re-randomized to REGN910-3 (6:2mg) Q8 and Q12) | 0 (Out of 148 that completed Week 12,143 re-randomized to Aflibercept 2mg Q8, Q12, REGN910-3 (6:2mg) Q8) | 44 (Out of 96 that were re-randomized, 44 re-randomized from REGN910-3(6:2 mg)Q4 to REGN910-3(6:2 mg)Q8) | 52 (Out of 96 that were re-randomized, 52 re-randomized from REGN910-3(6:2 mg)Q4 to REGN910-3(6:2 mg)Q12) | 46 (Out of 143 that were re-randomized, 46 re-randomized from Aflibercept 2mg Q4 to Aflibercept 2mg Q8) | 48 (Out of 143 that were re-randomized, 48 re-randomized from Aflibercept 2mg Q4 to Aflibercept 2mg Q12) | 49 (Out of 143 that were re-randomized, 49 re-randomized from Aflibercept 2mg Q4 to REGN910-3 (6:2mg) Q8)
Completed | 44 | 0 | 0 | 42 | 50 | 46 | 43 | 45
Not Completed | 1 | 0 | 0 | 2 | 2 | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- REGN910-3 (6 mg:2 mg): Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, week 4 and week 8 for 3 initial doses. At week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) at week 16 or Week 20 and Q8 or Q12 through week 32.
- Aflibercept 2 mg: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At week 12, participants were re-randomized to receive IAI or REGN910-3 (6 mg:2 mg) at week 16 or 20 and Q8 through week 32.
- Total: Total of all reporting groups
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg | Total
Number analyzed (Participants) | 50 | 100 | 152 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (9.12) | 62.5 (10.36) | 59.5 (10.20) | 61.0 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 49 | 68 | 138
  Male | 29 | 51 | 84 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 21 | 26 | 53
  Not Hispanic or Latino | 44 | 78 | 125 | 247
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 3 | 4
  Asian | 1 | 2 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 11 | 8 | 19 | 38
  White | 37 | 87 | 121 | 245
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 12
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. Best Corrected Visual Acuity (BCVA) score was measured using an eye chart and was reported as the number of letters read correctly at a testing distance of 4 meters using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Change from baseline calculated by subtracting baseline value from observed post-baseline value at Week 12.
Time Frame: Baseline, Week 12
Population: Full analysis set included all randomized participants who received any study drug, had baseline measurement of BCVA & at least 1 post-baseline assessment of BCVA. Last observation carried forward (LOCF) method was used to impute missing data. Here "Overall Number of Participants Analyzed" = Participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg
Number analyzed (Participants) | 47 | 99 | 150
Letters correctly read | 6.8 (7.30) | 8.5 (6.89) | 8.8 (9.71)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg: 2 mg) vs Aflibercept 2 mg; Test type: Superiority — Analysis was performed using analysis of covariance (ANCOVA) model with baseline measurement as a covariate and treatment group as fixed factors; p = 0.1368, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -2.09, 95% CI 2-sided [- 4.84 to 0.67]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept 2 mg; Analysis was performed using analysis of covariance (ANCOVA) model with baseline measurement as a covariate and treatment group as fixed factors; Test type: Superiority; p = 0.9716, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.04, 95% CI 2-sided [- 2.10 to 2.18]

2. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 36
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. BCVA score was measured using an eye chart and was reported as the number of letters read correctly at a testing distance of 4 meters using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Change from baseline calculated by subtracting baseline value from observed post-baseline value at Week 36.
Time Frame: Baseline, Week 36
Population: FAS secondary randomization set = all participants in full analysis set (FAS) who had completed study through week 12, received any study drug after secondary randomization or after Week 12, had BCVA assessment at Week 12 & had at least 1 post-Week 16 BCVA assessment. Overall Number of Participants Analyzed=Participants evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 45 | 44 | 52 | 46 | 48 | 49
Letters correctly read | 9.8 (9.92) | 10.3 (8.20) | 8.5 (7.74) | 8.7 (10.65) | 10.0 (10.37) | 11.9 (12.01)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg: 2 mg) vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; Analysis was performed using ANCOVA model with baseline measurement as a covariate, and treatment group and BCVA stratification variable as fixed factors; Test type: Superiority; p = 0.1665, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 2.15, 95% CI 2-sided [-0.90 to 5.20]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2223, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 1.90, 95% CI 2-sided [-1.16 to 4.95]
Statistical Analysis 3: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7943, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.39, 95% CI 2-sided [-2.54 to 3.32]
Statistical Analysis 4: Comparison: Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6655, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.66, 95% CI 2-sided [-2.35 to 3.67]
Statistical Analysis 5: Comparison: Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 vs Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1278, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 2.33, 95% CI 2-sided [-0.67 to 5.33]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3159, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -1.51, -1.51% CI 2-sided [-4.47 to 1.45]
Statistical Analysis 7: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8537, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.27, 95% CI 2-sided [-3.18 to 2.63]

3. Secondary Outcome: Change From Baseline in Central Sub-field Retinal Thickness (CST) Measured by Spectral Domain Optical Coherence Tomography (SD-OCT) at Week 12
Description: Central Sub-field Retinal Thickness (CST) was assessed using Spectral Domain Optical Coherence Tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from baseline indicated improvement. Change from baseline calculated by subtracting baseline value from LOCF post-baseline value at Week 12.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg
Number analyzed (Participants) | 46 | 99 | 150
Microns | -169.4 (155.86) | -184.0 (143.69) | -174.6 (160.36)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg: 2 mg) vs Aflibercept 2 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.1105, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -24.43, 95% CI 2-sided [-54.46 to 5.61]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept 2 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0183, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -27.79, 95% CI 2-sided [- 50.83 to - 4.74]

4. Secondary Outcome: Change From Baseline in Central Sub-field Retinal Thickness (CST) Measured by Spectral Domain Optical Coherence Tomography (SD-OCT) at Week 36
Description: CST was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from baseline indicated improvement. Change from baseline calculated by subtracting baseline value from LOCF post-baseline value at Week 36.
Time Frame: Baseline, Week 36
Population: FAS secondary randomization set was used. Here "Overall Number of Participants Analyzed"= Participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 44 | 44 | 52 | 46 | 48 | 49
Microns | -210.4 (164.06) | -223.4 (145.35) | -193.7 (158.29) | -161.9 (125.99) | -210.6 (202.15) | -203.7 (163.08)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg: 2 mg) vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0040, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -55.91, 95% CI 2-sided [- 93.81 to - 18.01]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0365, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -40.51, 95% CI 2-sided [-78.46 to -2.57]
Statistical Analysis 3: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0454, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -37.15, 95% CI 2-sided [-73.53 to -0.77]
Statistical Analysis 4: Comparison: Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9266, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 1.75, 95% CI 2-sided [-35.54 to 39.03]
Statistical Analysis 5: Comparison: Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 vs Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4116, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -15.49, 95% CI 2-sided [-52.58 to 21.59]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8574, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 3.36, 95% CI 2-sided [-33.42 to 40.14]
Statistical Analysis 7: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0351, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -38.90, 95% CI 2-sided [-75.06 to -2.73]

5. Secondary Outcome: Percentage of Participants With a ≥ 2-step Improvement at Week 12 in Diabetic Retinopathy Severity Scale (DRSS) From Baseline
Description: The Diabetic Retinopathy Disease Severity Scale (DRSS) was used to describe overall retinopathy severity. It measured the 5 levels of diabetic retinopathy ranging from absence of retinopathy to severe retinopathy (none, mild, moderate, severe, and proliferative).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg
Number analyzed (Participants) | 45 | 94 | 145
Percentage of participants | 13.3 | 21.3 | 15.2
Statistical Analysis 1: Comparison: REGN910-3 (3 mg: 2 mg) vs Aflibercept 2 mg; Analysis was performed using analysis of Cochran-Mantel-Haenszel model; Test type: Superiority; p = 0.7617, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = -1.8, 95% CI 2-sided [-13.5 to 9.8]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept 2 mg; Analysis was performed using analysis of Cochran-Mantel-Haenszel model; Test type: Superiority; p = 0.2268, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 6.1, 95% CI 2-sided [- 4.1 to 16.3]

6. Secondary Outcome: Percentage of Participants With a ≥ 2-step Improvement at Week 36 in Diabetic Retinopathy Severity Scale (DRSS) From Baseline
Description: as for outcome 5
Time Frame: Baseline, Week 36
Population: FAS secondary randomization set was used. Overall Number of Participants Analyzed = Participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 45 | 44 | 50 | 46 | 47 | 48
Percentage of participants | 26.7 | 34.1 | 34.0 | 26.1 | 25.5 | 35.4
Statistical Analysis 1: Comparison: REGN910-3 (3 mg: 2 mg) vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; Difference with Confidence Interval was calculated using Mantel-Haenszel weighting scheme adjusted by BCVA stratification variable; Test type: Superiority; p = 0.8896, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = -1.3, 95% CI 2-sided [-20.4 to 17.7]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.5021, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 6.4, 95% CI 2-sided [-12.6 to 25.5]
Statistical Analysis 3: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.5273, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 6.0, 95% CI 2-sided [-12.8 to 24.7]
Statistical Analysis 4: Comparison: Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.8683, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = -1.5, 95% CI 2-sided [-19.7 to 16.6]
Statistical Analysis 5: Comparison: Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 vs Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3546, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 8.8, 95% CI 2-sided [-9.8 to 27.4]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.9801, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 0.2, 95% CI 2-sided [-19.0 to 19.5]
Statistical Analysis 7: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3528, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; difference in percentages = 8.8, 95% CI 2-sided [-9.9 to 27.4]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 36) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (Baseline up to Week 36).
Arm/Group | REGN910-3 (3 mg: 2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg
All-Cause Mortality (participants affected / at risk) | 5/50 | 0/100 | 4/152
Serious Adverse Events (participants affected / at risk) | 6/50 | 18/100 | 31/152
Other Adverse Events (participants affected / at risk) | 18/50 | 42/100 | 55/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN910-3 (3 mg: 2 mg) (N=50) | REGN910-3 (6 mg:2 mg) (N=100) | Aflibercept 2 mg (N=152)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal varices (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastric infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN910-3 (3 mg: 2 mg) (N=50) | REGN910-3 (6 mg:2 mg) (N=100) | Aflibercept 2 mg (N=152)
Conjunctival haemorrhage (Eye disorders) | 5 (6) | 3 (4) | 13 (16)
Dry eye (Eye disorders) | 0 (0) | 5 (5) | 1 (1)
Eye pain (Eye disorders) | 3 (4) | 3 (3) | 4 (4)
Vitreous detachment (Eye disorders) | 1 (1) | 8 (10) | 8 (8)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (7) | 7 (8)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (4) | 5 (6)
Blood pressure increased (Investigations) | 2 (2) | 7 (8) | 10 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 14 (15) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT02712008/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT02712008/SAP_001.pdf